CLINICAL TRIAL: NCT02484768
Title: A Phase II, Six-week, Randomised, Comparative, Double-blind Study of Intravenous Iron Isomaltoside 1000 Versus Placebo in Subjects With Restless Leg Syndrome With a 3 Month Extension
Brief Title: IV Iron Treatment of Restless Legs Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: as per GCP sponsor/company decision
Sponsor: Pharmacosmos A/S (Industry)
Collaborators: BioStata (Industry); Laboratory Corporation of America (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P-RLS-01
Record Dates: First submitted 2015-03-30; First posted 2015-06-30 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — iron isomaltoside 1000; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Infusion of 1000 mg iron isomaltoside 1000 at baseline. The infusion is diluted in 100 mL 0.9 % sodium chloride and given over approximately 15 min
  Interventions: Drug: Iron isomaltoside 1000
- Group B (Placebo Comparator): Infusion of 100 mL 0.9 % sodium chloride at baseline given over approximately 15 min
  Interventions: Drug: Sodium Chloride 0.9%

INTERVENTIONS:
Drug: Iron isomaltoside 1000 — Intravenous treatment
  Other Names: Monofer
  Arms: Group A
Drug: Sodium Chloride 0.9% — Intravenous treatment
  Arms: Group B

SUMMARY:
The purpose of this study is to to establish proof-of-concept for efficacy of iron isomaltoside 1000 in subjects with Restless Legs Syndrome.

The study is a randomised, comparative, double-blind study with a 3 months extension. Subjects with restless leg syndrome (RLS) will be randomised 2:1 to one of the following treat-ment groups:

* Group A (42 subjects): 1000 mg iron isomaltoside 1000
* Group B (21 subjects): Placebo infusion

Furthermore, non-responders, who continue to meet entry requirements, will receive 1000 mg iron isomaltoside 1000 at week 6.

DETAILED DESCRIPTION:
RLS is a disorder of sensation with a prevalence of around 2-5 % of the population. RLS is extremely responsive to dopaminergic agents, but a second issue is that iron deficiency states may precipitate RLS in as much as 25-30 % of subjects with iron deficiency. RLS appears to be related to deficits in brain iron content and metabolism. Magnetic resonance imaging (MRI) images demonstrate a decrease in substantia nigra and red nucleus iron content. The severity of this decrease in brain iron content is correlated with the severity of symptoms. A number of patients are quite resistant to dietary iron repletion but do resolve symptoms with high doses of intravenous (IV) iron.

For the individual subject, there will be 4 phases to the study which includes teleconferences (TCs) and 2 visits.

The treatment and treatment evaluation is the main study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Diagnosis of RLS based upon the CH-RLSq and HTDI
3. IRLS score ≥ 15 at baseline evaluation when off RLS medications
4. Willingness to participate and signing the informed consent form

Exclusion Criteria:

1. S-ferritin > 300 ng/mL and/or TfS > 50 %
2. Iron overload or disturbances in utilisation of iron (e.g. haemochromatosis and haemo-siderosis)
3. Known hypersensitivity to IV iron or any excipients in the investigational drug prod-ucts
4. Pregnant or nursing women. In order to avoid pregnancy, women of childbearing po-tential have to use adequate contraception (e.g. intrauterine devices, hormonal contra-ceptives, or double barrier method) during the whole study period and 7 days after the last dosing
5. History of active asthma within the last 5 years
6. Decompensated liver cirrhosis or active hepatitis (defined as ASAT or ALAT > 3 times upper limit of normal)
7. Active acute or chronic infections (assessed by clinical judgement supplied with WBC and CRP)
8. Rheumatoid arthritis with symptoms or signs of active inflammation
9. Pregnant or nursing women
10. Previous IV iron treatment for RLS
11. IV iron treatment within 1 year prior to screening
12. Blood transfusion within 4 weeks prior to screening
13. Planned elective surgery during the study
14. Participation in any other interventional study where the study drug has not passed 5 half-lives prior to the screening
15. Any other medical condition that, in the opinion of the Investigator, may cause the subject to be unsuitable for the completion of the study or place the subject at potential risk from being in the study, e.g. history of multiple allergies, a malignancy, uncon-trolled hypertension, unstable ischaemic heart disease, or uncontrolled diabetes melli-tus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
To measure the change in RLS symptoms from baseline to week 6 measured by the clinical global impression (CGI) score | 6 weeks

SECONDARY OUTCOMES:
Change in RLS symptoms from baseline to week 4 and month 2 and 3 measured by the CGI score | 3 months
Change in RLS symptoms from baseline to week 4 and 6 and month 2 and 3 measured by the International Restless Legs Scale (IRLS) | from baseline to t = 12 weeks
Time from baseline to start of RLS medication | from baseline to t = 6 weeks
Time from baseline to start of RLS medication or non-response (CGI ≥ 3 at week 6) | from baseline to t = 6 weeks

OTHER OUTCOMES:
Type and incidence of adverse drug reactions (ADRs) | from baseline to t = 18 weeks
Number of adverse events (AEs) of special interest | from baseline to t = 18 weeks
  (i.e. hypersensitivity symptoms such as: urticaria, oedema, bronchospasm, hypotension, cardiorespiratory arrest, syn-cope, unresponsiveness, or loss of consciousness at pre-specified time points in relation to administration of study drug)
Change in haematology parameters, s-sodium, s-potassium, s-calcium, s-phosphate, s-urea, s-creatinine, s-albumin, s-bilirubin, aspartate aminotransferase (ASAT), and ala-nine aminotransferase (ALAT) from baseline to week 6 and month 3 | from baseline to t = 18 weeks
Change in vital signs (heart rate and blood pressure) during drug administration | from baseline to t = 18 weeks
Clinical significant electrocardiogram (ECG) during drug administration | from baseline to t = 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard Allen, Assoc Prof, Principal Investigator — Johns Hopkins University Asthma& Allergy Bldg 1B76b 5501 Hopkins Bayview Blvd Baltimore, MD 21224 USA